CLINICAL TRIAL: NCT02583100
Title: Improving Outcomes in Cleft Palate Surgery Through an Audit and Feedback Intervention Directed at Surgeons
Brief Title: Improving Outcomes in Cleft Palate Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-5428
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Feedback (Experimental): Participants in this arm will receive intensive feedback on their complication rates, surgical technique, and peri-operative surgical management from peer surgeons participating in the study.
  Interventions: Behavioral: Intensive Feedback
- Routine Feedback (Active Comparator): Participants in this arm will receive routine feedback on their complication rates.
  Interventions: Behavioral: Routine Feedback

INTERVENTIONS:
Behavioral: Intensive Feedback — (1) receive feedback regarding their individual fistula rate and those of all other participants in the trial, (2) receive an analysis of their video-recorded operative technique by surgeon peers, (3) directly observe a peer surgeon with lower fistula rate, and (4) develop a personalized action plan with a target for improvement.
  Arms: Intensive Feedback
Behavioral: Routine Feedback — (1) receive feedback regarding their individual fistula rate and those of all other participants in the trial
  Arms: Routine Feedback

SUMMARY:
This is a pilot study to determine if an audit and feedback intervention decreases complication rates after cleft palate surgery.

DETAILED DESCRIPTION:
This study will determine whether a surgeon-directed audit and feedback intervention reduces rates of oro-nasal fistula after cleft palate repair. Fistula is an important potential complication of cleft palate repair.

The study also evaluates feasibility of standardized outcome measurement in the care of children with cleft lip and palate, acceptability of standardized measurement, and acceptability of the audit and feedback intervention among surgeons.

The results of this research will improve child health by enabling cleft surgeons to critically evaluate and improve their patient's outcomes.

ELIGIBILITY:
Inclusion Criteria:

Active surgeon performing cleft palate repair in the US or Canada.

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Oro-nasal Fistula | 12 weeks
  Presence or absence of fistula of the palate

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Grossoehme, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Thomas Sitzman, MD, Study Director — Phoenix Children's Hospital
Locations (6):
- United States (5):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Duke Children's Hospital, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Penn State Hershey Craniofacial Clinic, Hershey, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada